CLINICAL TRIAL: NCT05402813
Title: Longitudinal Study of the Natural History of Two Autosomal Recessive Non Syndromic Deafness (DFNB1A and DFNB9) in Children Up to 16 Years of Age
Brief Title: Natural History in Children Up to 16 Years with Mild to Profound Hearing Loss Due to Mutations in GJB2 / OTOF Genes
Acronym: Otoconex
Status: Recruiting | Type: Observational
Sponsor: Sensorion (Industry)
Responsible Party: Sponsor
Other Study IDs: SENS-NH01
Record Dates: First submitted 2022-05-16; First posted 2022-06-02 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Sensorineural Hearing Loss, Bilateral; AUNB1; DFNB1A; Congenital Deafness; DFNB9; OTOF Gene Mutation; GJB2 Gene Mutation
MeSH Terms: conditions — Hearing Loss, Sensorineural; Deafness, Autosomal Recessive 1A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1a: Patients without Cochlear Implant, with or without Hearing Aid(s) at study entry
  Interventions: Other: Pure Tone Audiometry Assessment; Other: Quality of Life Questionnaires
- Cohort 1b: Patients receiving unilateral or bilateral Cochlear Implant(s) during the study period, after study entry
  Interventions: Other: Pure Tone Audiometry Assessment; Other: Quality of Life Questionnaires
- Cohort 2: Patients with Cochlear Implant(s) (unilateral or bilateral) at study entry
  Interventions: Other: Pure Tone Audiometry Assessment; Other: Quality of Life Questionnaires

INTERVENTIONS:
Other: Pure Tone Audiometry Assessment — Collection of Pure Tone Audiometry data performed in routine practice during study period
Other: Quality of Life Questionnaires — Collection of Quality of Life questionnaire's answers during study period

SUMMARY:
The purpose of this study is to follow the natural history of non-syndromic hearing loss caused by mutations in two genes (GJB2 or OTOF) in children up to 16 years of age.

DETAILED DESCRIPTION:
The study aims to:

* better describe the prevalence of cases of DFNB1A and DFNB9, including the type of mutations, and to assess the clinical course of the disease in children up to 16 years of age who have a mild to profound deafness.
* better understand the audiological and genetic characteristics of the participants with congenital versus evolutive DFNB1A and DFNB9 deafness.

ELIGIBILITY:
Main Inclusion Criteria:

Participants meeting all the following main inclusion criteria will be eligible to participate in the study:

* Aged ≤ 16 years on the date of signed informed consent for cohort 1 and ≤ 10 years for cohort 2;
* With a diagnosis of non-syndromic, bilateral, mild to profound, sensorineural hearing loss (according to the American Speech Language-Hearing Association);
* With documented genotyping results showing mutation(s) in GJB2 or OTOF genes;
* Written informed consent as required by local regulations.
* Either without Cochlear Implant, or with unilateral or bilateral Cochlear Implant(s)

Exclusion Criteria:

Participants presenting with any of the following main exclusion criteria will not be included in the study

* Other type of deafness, such as unilateral deafness, persistent conductive deafness, malformation syndrome, syndromic deafness, known familial deafness linked to mutations in other genes than OTOF or GJB2;
* Documented genotyping results showing pathogenic mutation(s) in other gene(s) than GJB2 or OTOF genes in the tested panel;
* Unable and/or unwilling to comply with all the protocol requirements and/or study procedures.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male and female participants aged ≤ 16 years at selection, with a diagnosis of bilateral, moderate to profound, sensorineural, non-syndromic hearing loss, with genotyping results showing mutation(s) in GJB2 or OTOF genes, with and without cochlear implant (CI).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2028-11-18 (Estimated); Study Completion 2028-11-18 (Estimated)

PRIMARY OUTCOMES:
Audiological characteristics | Up to 4 years
  Pure Tone Audiometry, thresholds on 500, 1000, 2000, 4000 Hz Speech audiometry
Electrophysiological characteristics: ABR | Up to 4 years
  Auditory Brainstem Response, thresholds
Electrophysiological characteristics: OAE | Up to 4 years
  Otoacoustic Emissions thresholds

SECONDARY OUTCOMES:
Genotypic and phenotypic characterisation | 1 Day
  Genotypic and phenotypic characterisation of the population will be assessed in Cohort 1a.
  Frequency of autosomal recessive 1 and 9 deafness (GJB2 and OTOF genes) and type of mutations will be evaluated among the screened population of male and female children aged ≤ 10 years, with a diagnosis of bilateral moderate to profound, sensorineural, non-syndromic hearing loss.
Hearing-related Quality of Life questionnaire | Up to 4 years
  The Hearing Environments And Reflection on Quality of Life (HEAR-QL) measurement questionnaires will be used to assess the quality of life of children.
  Depending on child's age, the HEAR-QL questionnaires will be completed either by parents/caregivers (child aged 2 to 6 years) either by the child (child aged 7 to 12 years).
  The items of the questionnaires are focused on situations affecting interactions with family and friends, participation in social and school activities, and impact of Hearing Loss on the child's emotional well being.
  Children/parents will be asked to rate how frequently each item was a problem for them/child in the past month using the following response choices: "never" (1), "almost never" (2), "sometimes" (3), "often" (4), or "Almost always" (5). Scores are transformed with 1=100, 2=75, 3=50, 4=25, and 5=0 points. Higher scores indicate higher perceived Quality Of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie LOUNDON, MD, Principal Investigator — Necker Hospital
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No